CLINICAL TRIAL: NCT01856634
Title: Phase 1, Open-label, Multiple-dose, and Age De-escalation Trial to Assess the Pharmacokinetics, Safety and Tolerability of Delamanid (OPC 67683) in Pediatric Multidrug-resistant Tuberculosis Patients on Therapy With an Optimized Background Regimen of Anti-tuberculosis Drugs
Brief Title: Pharmacokinetic and Safety Trial to Determine the Appropriate Dose for Pediatric Patients With Multidrug Resistant Tuberculosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 242-12-232
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Multidrug Resistant Tuberculosis; Pediatric
Keywords: Tuberculosis; Tuberculosis, Multidrug-Resistant; Mycobacterium Infections; Actinomycetales Infections; Gram-Positive Infections; Bacterial Infections; Pediatric
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis; Mycobacterium Infections; Actinomycetales Infections; Bacterial Infections | interventions — OPC-67683

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: 12 to 17 years of age (Experimental): Group 1: 100 mg Delamanid BID for 10 days + OBR
  Interventions: Drug: 100 mg Delamanid; Drug: Optimized Background Regimen
- Group 2: 6 to 11 years of age (Experimental): 50 mg Delamanid BID for 10 days + OBR
  Interventions: Drug: 50 mg Delamanid; Drug: Optimized Background Regimen
- Group 3: 3 to 5 years of age (Experimental): 25 mg Pediatric Formulation Delamanid BID for 10 days + OBR
  Interventions: Drug: 25 mg Pediatric Formulation Delamanid; Drug: Optimized Background Regimen
- Group 4: Birth to 2 years of age (Experimental): Delamanid Pediatric Formulation (DPF) for 10 days + OBR. DPF dose based on patient's body weight during baseline visit:
  * Patient's > 10 kg will receive DPF 10 mg BID + OBR
  * Patient's > 8 kg and ≤ 10 kg will receive DPF 5 mg BID + OBR
  * Patients ≤ 8 kg will receive DPF 5 mg QD + OBR
  Interventions: Drug: 10 mg Delamanid Pediatric Formulation; Drug: 5 mg Delamanid Pediatric Formulation; Drug: Optimized Background Regimen

INTERVENTIONS:
Drug: 100 mg Delamanid — 100 mg Delamanid BID for 10 days
  Other Names: OPC-67683
  Arms: Group 1: 12 to 17 years of age
Drug: 50 mg Delamanid — 50 mg Delamanid BID for 10 days
  Other Names: OPC-67683
  Arms: Group 2: 6 to 11 years of age
Drug: 25 mg Pediatric Formulation Delamanid — 25 mg Pediatric Formulation Delamanid BID for 10 days
  Other Names: DPF
  Arms: Group 3: 3 to 5 years of age
Drug: 10 mg Delamanid Pediatric Formulation — Patients > 10 kg will receive DPF 10 mg BID for 10 days
  Other Names: DPF
  Arms: Group 4: Birth to 2 years of age
Drug: 5 mg Delamanid Pediatric Formulation — Patients > 8 kg and ≤ 10 kg will receive DPF 5 mg BID for 10 days
  Patients ≤ 8 kg will receive DPF 5 mg QD for 10 days
  Other Names: DPF
  Arms: Group 4: Birth to 2 years of age
Drug: Optimized Background Regimen — Selection and administration of the treatment medications (i.e. OBRs) will be based on WHO's Guidelines for the programmatic management of drug-resistant TB, in conjunction with national TB program guidelines in each country
  Other Names: OBR

SUMMARY:
The purpose of this trial is to determine the pediatric dose of delamanid that is equivalent to the adult dose already shown to be effective against multidrug-resistant tuberculosis.

DETAILED DESCRIPTION:
This trial will investigate the pharmacokinetics (PK) and safety of delamanid administered for 10 days to pediatric patients aged birth to 17 years who are also on therapy with an optimized background regimen. The purpose of the trial is to determine which dose in pediatric MDR-TB patients will result in delamanid plasma exposure similar to efficacious plasma exposure in adult MDR-TB patients. This is an age de-escalation trial in four groups:

Group 1: 12 to 17 years (100 mg BID; n=6) Group 2: 6 to 11 years (50 mg BID; n=6) Group 3: 3 to 5 years (25 mg BID; n=12) Group 4: Birth to 2 years (Dose based on patient's body weight, n=12)

* Patients > 10 kg will receive 10 mg BID
* Patients > 8 kg and ≤ 10 kg will receive 5 mg BID
* Patient ≤ to 8 kg will receive 5 mg QD

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MDR-TB OR
* Presumptive diagnosis of MDR-TB including one of the following:

  * Clinical specimen suggestive of TB
  * Persistent cough lasting > 2 weeks
  * Fever, weight loss, and failure to thrive
  * Findings on recent chest radiograph (prior to Visit 1) consistent with TB AND
  * Household contact of a person with known MDR-TB or a person who died while appropriately taking drugs for sensitive TB OR
  * On first-line TB treatment but with no clinical improvement
* Negative urine pregnancy test for female patients who have reached menarche
* Written informed consent/assent

Exclusion Criteria:

* Laboratory evidence of active hepatitis B or C
* Children with body weight < 5.5 kg
* For patients with HIV co-infection, CD4 cell count ≤ 1000/mm3 for children 1-5 years old, and ≤ 1500/mm3 for children less than 1 year old
* History of allergy to metronidazole and any disease or condition in which metronidazole is required
* Use of amiodarone within 12 months or use of other predefined antiarrhythmic medications within 30 days prior to first dose of delamanid
* Serious concomitant conditions
* Preexisting cardiac conditions
* Abnormalities in Screening ECG (including AV block, BBB or hemi-block, QRS prolongation > 120 msec, or QTcF > 450 msec in both males and females)
* Concomitant condition such as renal impairment characterized by serum creatinine levels >1.5 mg/dL, hepatic impairment (ALT or AST > 3x ULN), or hyperbilirubinemia characterized by total bilirubin > 2x ULN
* Current diagnosis of severe malnutrition or kwashiorkor
* Positive urine drug screen (Groups 1 and 2 only)
* Rifampicin and/or moxifloxacin within 1 week prior to the first dose of delamanid and/or any prior or concurrent use of bedaquiline
* Lansky Play Performance Score < 50 (not applicable for children < 1 year old) or Karnofsky Score < 50
* Administered an IMP within 1 month prior to Visit 1
* Pregnant, breast-feeding, or planning to conceive or father a child within the timeframe described in the information consent form (Groups 1 and 2 only)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations | Days 1, 2, 10, 11, 13 (Groups 1 and 2 only), 15, 18
  Plasma concentrations (Cmax, tmax, AUC 0-24h, accumulation ratio, apparent terminal elimination half-life, apparent total clearance) of delamanid and its metabolites on Days 1, 2, 10, 11, 13 (Groups 1 and 2 only), 15, 18.

SECONDARY OUTCOMES:
Adverse Events | 40 Days
  Number of reported adverse events
Safety Summary | 40 Days
  Summary statistics of subjects with clinically significant abnormal laboratory test results, vitals, ECGs
Palatability of the Pediatric Formulation | Days 1 and 10
  Palatability of the pediatric formulation will be assessed using an age-appropriate visual hedonic scale and clinical assessment for Groups 3 and 4 only.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hafkin, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (2):
- De La Salle Health Sciences Institute, Dasmariñas, Cavite, Philippines
- Brooklyn Chest Hospital, Ysterplaat, Cape Town, South Africa

REFERENCES:
- [Derived] Garcia-Prats AJ, Frias M, van der Laan L, De Leon A, Gler MT, Schaaf HS, Hesseling AC, Malikaarjun S, Hafkin J. Delamanid Added to an Optimized Background Regimen in Children with Multidrug-Resistant Tuberculosis: Results of a Phase I/II Clinical Trial. Antimicrob Agents Chemother. 2022 May 17;66(5):e0214421. doi: 10.1128/aac.02144-21. Epub 2022 Apr 11. PMID 35404075